CLINICAL TRIAL: NCT03003000
Title: A Randomized, Placebo- and Active-controlled Multi-country, Multi-centre Parallel Group Study to Evaluate the Efficacy and Safety of a Fixed Dose Combination of 400 mg Ibuprofen and 100 mg Caffeine Compared to Ibuprofen 400 mg and Placebo in Patients With Acute Lower Back or Neck Pain.
Brief Title: Ibuprofen/Caffeine Lower Back or Neck Pain Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1335.5; 2016-000902-12 (EudraCT Number)
Record Dates: First submitted 2016-11-17; First posted 2016-12-26 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Back Pain; Neck Pain
MeSH Terms: conditions — Back Pain; Neck Pain | interventions — Ibuprofen; Caffeine

ARMS (3):
- ibuprofen + caffeine (Experimental): Fixed Dose Combination
  Interventions: Drug: ibuprofen; Drug: caffeine
- ibuprofen (Active Comparator)
  Interventions: Drug: ibuprofen
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ibuprofen
  Arms: ibuprofen; ibuprofen + caffeine
Drug: caffeine
  Arms: ibuprofen + caffeine
Drug: placebo
  Arms: placebo

SUMMARY:
To assess the efficacy and safety of a 400 mg ibuprofen/100 mg caffeine tablet in comparison to a 400 mg ibuprofen tablet for the treatment of acute lower back or neck pain. To assess the safety and tolerability of a 400 mg ibuprofen/100 mg caffeine tablet in comparison to a 400 mg ibuprofen tablet and a placebo tablet.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent at Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation.
* Male or female patients who are >=18 years with current diagnosis of acute back pain or of neck pain for at least 24 hours, but less than 21 days.
* Acute back pain or acute neck pain resulting in Pain on Movement (POM) >=5 on the 0-10 Numerical Rating Scale (NRS) for at least one POM procedure out of 5 standardised procedures.
* Sensitivity to algometric pressure on the painful trigger point <= 25 N/cm².
* Women of childbearing potential must be ready and able to use highly effective methods of birth control.
* Reliable, cooperative, and of adequate intelligence to record the requested information on the analgesic questionnaires.
* Examined by the attending physician and medically cleared to participate in the study
* In good general health, with a body mass index (BMI) < 30, and have no contraindications to any of the study medication

Exclusion criteria:

* History of 3 or more episodes of back or neck pain in the last 6 months excluding the current episode.
* Patients with pain at rest >= 9
* Patient with chronic back or neck pain as defined as pain for 3 weeks or longer.
* Back or neck pain that is attributable to any identifiable cause (eg. disc prolapse, spondylolisthesis, osteomalacia, inflammatory arthritis, metabolic, neurological diseases or tumour)
* Any strains of the back or neck muscles documented by clinical evaluation and anamnesis that occurred 21 days to 3 months prior to the screening visit.
* Surgery due to back or neck pain or rehabilitation due to back or neck pain in the last 12 months.
* Prior use within the last 3 days before Visit 1 or concomitant use of any anti- inflammatory drugs, heparinoids, muscle relaxants or analgesics (including but not limited to short-acting glucocorticoids, non-steroidal anti-inflammatory drugs [NSAIDs], herbal preparations) for the same indication or other indications.
* Spinal injections should have been discontinued in due time (investigator's judgment) before patient enrollment to allow complete wash-out of the active ingredient based on investigator's judgment.
* Known severe hepatocellular insufficiency, severe renal insufficiency or Gilbert's syndrome (Morbus Meulengracht)
* Patients taking Central Nervous System (CNS) or other psychotropic drugs, or any nutritional supplement known to have psychotropic effects such as St. John's Wort, Chapparal, Comfrey, Germander, Gin Bu Huan, Kava, Pennyroyal Skullcap, or Valerian within two months of taking the first dose of study medication. Patients who have been on stable doses of these medications for at least two months will be allowed into the study, as long as they maintain this dose throughout the study, and their condition is judged stable by the Principal Investigator
* Any other medical condition that would interfere with efficacy and safety assessments based on investigator's judgment or any on-going clinical condition that would jeopardize patient's or site personnel's safety or study compliance based on investigator judgment
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-09-24 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (18):
- Germany (15):
  - Dünnwaldpraxis, Köln, Cologne
  - Praxis Dr. Steinebach, Essen, Essen
  - Praxis Dr. Schaefer, 45355 Essen, Essen
  - Studienzentrum Bocholderstraße, Essen
  - Unterfrintroper Hausarztzentrum, Essen
  - Praxis Dr. Pabst, Gilching, Gilching
  - Praxis Kai Gastl, Gilching
  - medicoKIT GmbH, Goch
  - Clinical Research Dr. Martz, Hamburg
  - Praxis Dr. Dahmen, 22415 Hamburg, Hamburg
  - Praxis Dr. Chevts, 76199 Karlsruhe, Karlsruhe
  - Praxis Dr. Klein, Künzing, Künzing
  - Anästhesiologie Rheinbach, Rheinbach
  - Praxis Dr. Sauter, Wangen
  - Neurologie und Psychiatrie / Psychotherapie, Westerstede
- Russia (3):
  - State Healthcare Institution, City Out-Patient's Clinic #109, Saint Petersburg
  - Medical Centre "Reavita Med SPb" LLC, Saint Petersburg
  - City Outpatient dep.no.107;clinc.pharmacology,st.petersburg, Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo and active-controlled, double-blind, 3-arm, parallel trial, comparing the effect of the fixed dose combination of 400 milligram (mg) ibuprofen&100 mg caffeine versus 400 mg ibuprofen and placebo in patients with acute neck or back pain randomly assigned in 2:2:1 ratio respectively.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered/randomised to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Placebo: Patients were administered placebo matching ibuprofen and ibuprofen/caffeine film-coated tablets orally 3 times daily with intervals of 6 to 8 hours (while awake) on Day 1 until the morning of Day 6.
- Ibuprofen: Patients were administered film-coated tablets orally containing 400 mg ibuprofen 3 times daily with intervals of 6 to 8 hours (while awake) on Day 1 until the morning of Day 6.
- Ibuprofen and Caffeine: Patients were administered film-coated tablets orally containing 400 mg ibuprofen and 100 mg caffeine 3 times daily with intervals of 6 to 8 hours (while awake) on Day 1 until the morning of Day 6.
Period: Overall Study
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Started (Randomized and treated) | 126 | 253 | 256
Completed | 121 | 249 | 251
Not Completed | 5 | 4 | 5
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Non-compliant with protocol | 0 | 1 | 1
Not completed — Refused to continue medication | 2 | 0 | 0
Not completed — Other than listed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS comprised all randomised patients who took at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine | Total
Number analyzed (Participants) | 126 | 253 | 256 | 635
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: TS
  Years | 46.3 (15.00) | 45.5 (16.40) | 44.8 (17.00) | 45.4 (16.36)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: TS
  Participants
    Female | 75 | 155 | 143 | 373
    Male | 51 | 98 | 113 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for ethnicity data. Population: TS
  Participants
    Hispanic or Latino | 1 | 0 | 0 | 1
    Not Hispanic or Latino | 125 | 253 | 256 | 634
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for race data. Population: TS
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 0 | 1 | 3 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 3 | 2 | 5
    White | 125 | 249 | 251 | 625
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Pain on movement worst procedure score (0-10) [Mean (Standard Deviation); unit: Unit on scale] — POM was assessed by the patient at the performance of one standardized, muscle group specific movement and was measured by a numerical rating scale ranging from 0 = 'no pain'to 10 = 'worst pain possible for this condition'. Population: Treated Set
  Unit on scale | 6.9 (1.07) | 6.8 (1.15) | 6.6 (1.15) | 6.7 (1.14)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain on Movement (POM) With Regard to the Worst Procedure (WP) Between Baseline and Day 2 (Morning, 2 Hours After Drug Intake)
Description: The change in pain on movement (POM) with regard to the worst procedure (WP), i.e. the procedure with the highest pain score at baseline (POMwp), between baseline (morning of Day 1, pre-dosing) and Day 2 (morning, 2 hour (h) after drug intake).
  POM was assessed by the patient at the performance of one standardized, muscle group specific movement and was measured by a numerical rating scale ranging from 0 = 'no pain'to 10 = 'worst pain possible for this condition'.
  The procedure resulting in highest POM at baseline (worst procedure, POMWP) was repeated for an individual patient. If 2 or more procedures gave the same highest POM, the patient was asked which of the procedures giving the highest POM scores he/she considered the most unpleasant.
  Change in POMwp was calculated as baseline POMwp - POMwp at Day 2 - indicating a reduction in POMwp, where the result is positive.
Time Frame: Baseline and Day 2
Population: Full analysis set (FAS): FAS comprised all patients in the TS who provided a baseline value for POMWP at Visit 1 (before drug intake) and at least 1 POMWP post-treatment value at Visit 1 (Day 1 morning, 2 h after drug intake) and at Visit 2 (Day 2, morning, 2 h after drug intake).
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Number analyzed (Participants) | 126 | 253 | 256
Unit on scale | 1.712 (0.1422) | 1.998 (0.1042) | 1.869 (0.1030)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen and Caffeine; Superiority of ibuprofen and caffeine versus ibuprofen as well as ibuprofen and caffeine versus placebo had to be shown to reject the overall null hypothesis that there is no difference in change in POMWP between baseline and Day 2 (morning, 2 h after drug intake) between patients treated with ibuprofen/caffeine and patients treated with placebo; Test type: Superiority; p = 0.3446, Mixed effect Model Repeated Measurement — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; Mean Difference (Final Values) = 0.156, 95% CI 2-sided [-0.168 to 0.480] — Adjusted mean change from baseline ibuprofen and caffeine - Adjusted mean change from baseline placebo. A positive result favors the treatment with ibuprofen and caffeine; Mixed effect model for repeated measures analysis (MMRM) includes fixed, categorical effects of treatment, country, worst procedure site, time and interaction terms for treatment-by-time, treatment-by-stratum-by-time, treatment-by-stratum and stratum-by-time interaction, as well as the continuous fixed covariates of baseline POMwp and baseline-by-time interaction, using unstructured covariance matrix
Statistical Analysis 2: Comparison: Ibuprofen vs Ibuprofen and Caffeine; Superiority of ibuprofen and caffeine versus ibuprofen as well as ibuprofen and caffeine versus placebo had to be shown to reject the overall null hypothesis that there is no difference in change in POMWP between baseline and Day 2 (morning, 2 h after drug intake) between patients treated with ibuprofen/caffeine and patients treated with ibuprofen; Test type: Superiority; p = 0.3358, Mixed effect Model Repeat Measurement — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; Mean Difference (Final Values) = -0.129, 95% CI 2-sided [-0.392 to 0.134] — Adjusted mean change from baseline ibuprofen and caffeine - Adjusted mean change from baseline ibuprofen. A positive result favors the treatment with ibuprofen and caffeine; [other analysis details as in outcome 1, analysis 1]

2. Secondary Outcome: The Area Under the Curve (AUC) for Pain on Movement (POM) With Regard to the Worst Procedure (POMwp) Between Baseline and Day 4 (Morning) (POMwpAUC72hour (h))
Description: This is a key secondary endpoint. The area under the curve (AUC) for pain on movement (POM) with regard to the worst procedure (POMwp) between baseline and Day 4 (morning), (POMwpAUC72h ). POM was assessed by the patient at the performance of one standardized, muscle group specific movement and was measured by a numerical rating scale ranging from 0 = 'no pain'to 10 = 'worst pain possible for this condition'. A higher AUC value indicates higher POMwp
Time Frame: Baseline, Day 1, Day 2 and Day 4 (morning)
Population: Treated Set (TS): The TS comprised all randomised patients who took at least 1 dose of trial medication.
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Number analyzed (Participants) | 126 | 253 | 256
Unit on scale | 4.800 (0.1266) | 4.461 (0.0942) | 4.512 (0.0931)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.0474, ANCOVA — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; ANCOVA included treatment, country, and worst procedure site as fixed effects and baseline POMwp as a continuous covariate; Mean Difference (Final Values) = -0.288, 95% CI 2-sided [-0.572 to -0.003] — Adjusted mean ibuprofen and caffeine - Adjusted mean placebo. A negative result favors ibuprofen and caffeine
Statistical Analysis 2: Comparison: Ibuprofen vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.6658, ANCOVA — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; The ANCOVA included treatment, country, and worst procedure site as fixed effects and baseline POMwp as a continuous covariate; Mean Difference (Final Values) = 0.051, 95% CI 2-sided [-0.180 to 0.282] — Adjusted mean ibuprofen and caffeine - Adjusted mean ibuprofen. A negative result favors ibuprofen and caffeine

3. Secondary Outcome: The Area Under the Curve (AUC) for the Procedure With the Highest Pain Score at Baseline (POMWP) Between Baseline and Day 6 (Morning) (POM(WP)AUC(120h))
Description: This is a key secondary endpoint. The area under the curve for pain on movement with regard to the worst procedure between baseline and Day 6 (morning) (POM(WP)AUC(120h).
  POM was assessed by the patient at the performance of one standardized, muscle group specific movement and was measured by a numerical rating scale ranging from 0 = 'no pain'to 10 = 'worst pain possible for this condition'. A higher AUC value indicates higher POMwp.
Time Frame: Baseline, Day 1, Day 2, Day 4 and Day 6 (morning)
Population: TS
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Number analyzed (Participants) | 126 | 253 | 256
Unit on scale | 4.175 (0.1334) | 3.718 (0.0992) | 3.776 (0.0981)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.0091, ANCOVA — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.399, 95% CI 2-sided [-0.698 to -0.100] — Adjusted mean ibuprofen and caffeine - Adjusted mean placebo. A negative result favors ibuprofen and caffeine
Statistical Analysis 2: Comparison: Ibuprofen vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.6387, ANCOVA — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; [statistical method as in outcome 2, analysis 2]; Mean Difference (Final Values) = 0.058, 95% CI 2-sided [-0.185 to 0.302] — Adjusted mean ibuprofen and caffeine - Adjusted mean ibuprofen. A negative result favors ibuprofen and caffeine

4. Secondary Outcome: Change in Pressure Algometry Between Baseline and Day 2 (Morning, 2 Hour After Drug Intake)
Description: Change in pressure algometry between baseline and Day 2 (morning, 2 h after drug intake).
  Pressure algometry was determined by the investigator as the pressure value (N/cm2) at a defined trigger point which is located in the area of POMWP. The measurement was performed by using a Somedic Algometer (Somedic AB, Sweden) or an equivalent calibrated and certified device. The pain reaction was determined by placing the algometer on the trigger point, i.e. an area of 1 cm² for which the patient indicated most painful tenderness. The pressure was constantly increased until the patient asked not to increase the pressure anymore. Upon this pain reaction, the corresponding pressure value was documented in the Electronic case report form (eCRF). The trigger point was to be marked with a ball pen to be able to repeat the subsequent assessment at the same position. Change in pressure was calculated as baseline pressure - pressure at Day 2, with a negative result indicating an improvement.
Time Frame: Baseline and Day 2 (morning, 2 h after drug intake)
Population: TS
Measure: Least Squares Mean (Standard Error); unit: newton/centimeter² (N/cm^2)
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Number analyzed (Participants) | 126 | 253 | 256
newton/centimeter² (N/cm^2) | -3.734 (0.6107) | -3.331 (0.4396) | -3.175 (0.4366)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen and Caffeine; Mixed effect model for repeated measures (MMRM) includes fixed, categorical effects of treatment, country, worst procedure site, time and interaction terms for treatment-by-time as well as the continuous fixed covariates of baseline pressure algometry and baseline-by-time interaction, using unstructured covariance matrix; Test type: Superiority; p = 0.4398, Mixed effect model for repeated measures — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; Mean Difference (Final Values) = 0.559, 95% CI 2-sided [-0.861 to 1.979] — Adjusted mean change ibuprofen and caffeine - Adjusted mean change placebo. A negative result favors ibuprofen and caffeine
Statistical Analysis 2: Comparison: Ibuprofen vs Ibuprofen and Caffeine; MMRM includes fixed, categorical effects of treatment, country, worst procedure site, time and interaction terms for treatment-by-time as well as the continuous fixed covariates of baseline pressure algometry and baseline-by-time interaction, using unstructured covariance matrix; Test type: Superiority; p = 0.7911, Mixed effect Model Repeat Measurement — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; Mean Difference (Final Values) = 0.156, 95% CI 2-sided [-1.002 to 1.314] — Adjusted mean change ibuprofen and caffeine - Adjusted mean change ibuprofen. A negative result favors ibuprofen and caffeine

5. Secondary Outcome: Global Assessment of Efficacy by the Patient at the End of Treatment (Morning of Day 6)
Description: Global assessment of efficacy by the patient at the end of treatment (morning of Day 6) is presented. The patient/investigator assessed the overall efficacy of the trial treatment on a 4-point verbal rating scale by answering the question: "How would you rate the overall effect of the trial medication for relieving back or neck pain?" (0 = poor; 1 = fair; 2 = good; 3 = very good).
Time Frame: At the end of treatment (morning of Day 6)
Population: TS including participants with available data for global assessment of efficacy
Measure: Number; unit: Participants
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Number analyzed (Participants) | 123 | 253 | 255
Participants
  Very good | 14 | 43 | 41
  Good | 46 | 115 | 116
  Fair | 35 | 57 | 66
  Poor | 28 | 38 | 32
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.0045, Regression, Logistic — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; An ordinal logistic regression model adjusting for country and worst procedure site; Odds Ratio (OR) = 1.777, 95% CI 2-sided [1.195 to 2.642] — An odds ratio >1 indicates better efficacy for ibuprofen and caffeine than for the comparator
Statistical Analysis 2: Comparison: Ibuprofen vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.9603, Regression, Logistic — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; An ordinal logistic regression model adjusting for country and worst procedure site; Odds Ratio (OR) = 1.008, 95% CI 2-sided [0.732 to 1.389] — An odds ratio >1 indicates better efficacy for ibuprofen and caffeine than for the comparator

6. Secondary Outcome: Number of Patients With a Decrease in POMwp of at Least 30% or 50% Between Baseline and Day 2 (Morning, 2 h After Drug Intake)
Description: Number of patients with a decrease in POMwp of at least 30% or 50% between baseline and Day 2 (morning, 2 h after drug intake.
Time Frame: Baseline and Day 2 (morning, 2 h after drug intake)
Population: TS
Measure: Number; unit: Participants
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Number analyzed (Participants) | 126 | 253 | 256
Participants
  Patients with a decrease of ≥30% | 49 | 111 | 101
  Patients with a decrease of ≥50% | 17 | 59 | 44
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.9022, likelihood-ratio test — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; The likelihood-ratio test was used to test treatment differences for patients with a decrease of ≥30%; Odds Ratio (OR) = 1.028, 95% CI 2-sided [0.663 to 1.592] — An odds ratio >1 indicates better efficacy for ibuprofen and caffeine than for the comparator; Results are based on the Logistic regression. Logistic regression model was adjusted for the categorical covariates country and worst procedure site
Statistical Analysis 2: Comparison: Ibuprofen vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.3129, likelihood-ratio test — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; The likelihood-ratio test was used to test treatment differences for patients with a decrease of ≥30%; Odds Ratio (OR) = 0.834, 95% CI 2-sided [0.586 to 1.187] — An odds ratio >1 indicates better efficacy for ibuprofen and caffeine than for the comparator; [other analysis details as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.3301, likelihood-ratio test — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; The likelihood-ratio test was used to test treatment differences for patients with a decrease of ≥50%; Odds Ratio (OR) = 1.354, 95% CI 2-sided [0.736 to 2.494] — An odds ratio >1 indicates better efficacy for ibuprofen and caffeine than for the comparator; [other analysis details as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Ibuprofen vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.0864, likelihood-ratio test — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; The likelihood-ratio test was used to test treatment differences for patients with a decrease of ≥50%; Odds Ratio (OR) = 0.680, 95% CI 2-sided [0.437 to 1.057] — An odds ratio >1 indicates better efficacy for ibuprofen and caffeine than for the comparator; [other analysis details as in outcome 6, analysis 1]

7. Secondary Outcome: Time to First Meaningful POMwp Relief Within 2 h After the First Dose of Trial Medication
Description: Time to event analysis of patients with first meaningful POMwp relief within 2 h after the first dose of trial medication. The percentage of observed patients with a meaningful POMwp relief within 2 h after the first dose of trial medication was reported. The procedure which resulted in the highest POM at baseline (POMwp) was repeated by the investigator 10, 20, 30, 60 and 120 min after the first dose of trial medication. The POMwp relief score (POMwpRS) was assessed by the patient at each of these time points by using a 5-point verbal rating scale (0 = no POMwp relief; 1 = little or perceptible POMwp relief; 2 = meaningful POMwp relief; 3 = a lot of POMwp relief; 4 = complete POMwp relief).
  The time to first meaningful POMWP relief was the earliest assessment time point after the first application of the trial medication at which the patient reported a score of ≥2.
Time Frame: Within 2 h after the first dose of trial medication
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
Number analyzed (Participants) | 126 | 253 | 256
Percentage of participants
  0 to ≤10 min | 1.6 | 0.8 | 0.8
  >10 to ≤20 min | 1.6 | 2.0 | 1.2
  >20 to ≤30 min | 1.6 | 2.4 | 2.0
  >30 to ≤60 min | 5.6 | 9.1 | 5.5
  >60 to <=120 | 8.7 | 8.3 | 10.2
  >120 min | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.9384, Log Rank — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; p-value based on a stratified log-rank test
Statistical Analysis 2: Comparison: Ibuprofen vs Ibuprofen and Caffeine; Test type: Superiority; p = 0.3534, Log Rank — No adjustment for multiplicity issues was made for this comparison. The level of significance was 0.05; p-value based on a stratified log-rank test

ADVERSE EVENTS:
Time Frame: From first drug administration until 24 hour after last intake of trial medication, up to 7 days.
Description: Treated Set (TS) (The TS comprised all randomised patients who took at least 1 dose of trial medication) was used for adverse event reporting.
Arm/Group | Placebo | Ibuprofen | Ibuprofen and Caffeine
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/253 | 0/256
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/253 | 0/256
Other Adverse Events (participants affected / at risk) | 0/126 | 0/253 | 0/256

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT03003000/SAP_000.pdf
  • Study Protocol (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03003000/Prot_001.pdf